CLINICAL TRIAL: NCT06559696
Title: Internal Mammary Lymph Nodes Irradiation in High-risk Breast Cancer After Neoadjuvant Chemotherapy: a Phase III Randomized, Controlled Clinical Trial
Brief Title: Internal Mammary Lymph Nodes Irradiation in High-risk Breast Cancer After Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Yong Yang, M.D., Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMUUH-BC-2401
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Internal mammary nodal; Radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- internal mammary nodal irradiation (Experimental): chest wall/whole breast and supraclavicular+-axillary nodal plus internal mammary nodal irradiation
  Interventions: Radiation: internal mammary nodal irradiation
- No internal mammary node irradiation (Active Comparator): chest wall/whole breast and supraclavicular+-axillary nodal irradiation
  Interventions: Radiation: No internal mammary node irradiation

INTERVENTIONS:
Radiation: internal mammary nodal irradiation — chest wall/whole breast and supraclavicular +-axillary plus internal mammary nodal irradiation (50 Gy in 25 fractions or 40Gy in 15 fractions).
  Arms: internal mammary nodal irradiation
Radiation: No internal mammary node irradiation — chest wall/whole breast and supraclavicular +-axillary irradiation (50 Gy in 25 fractions or 40Gy in 15 fractions).
  Arms: No internal mammary node irradiation

SUMMARY:
The aim of this study is to explore the impact of internal mammary nodal irradiation on disease-free survival in high-risk breast cancer patients (ypN+or supra/subclavicular lymph node positive) after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a prospective, randomized phase 3 trial. Breast cancer patients with axillary lymph node-positive or supra/subclavicular lymph node metastasis underwent neoadjuvant chemotherapy were included. Patients underwent regional nodal irradiation along with breast or chest wall irradiation and randomly allocated to either IMNI or no IMNI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* Underwent neoadjuvant chemotherapy
* Eastern Cooperative Oncology Group Performance Status Scale 0-2
* ypN+ after neoadjuvant chemotherapy or supraclavicular/subclavicular lymph node metastasis before system therapy
* No distant metastases
* No internal mammary nodes metastases based on images before system therapy
* Willing to follow up
* Written,informed consent

Exclusion Criteria:

* Without neoadjuvant chemotherapy
* Distant metastases
* Simultaneous bilateral breast cancer
* Pathological confirmation or imaging consideration of lymph node metastasis in the internal mammary before system therapy
* Had simultaneous or previous secondary malignancies, except for non-malignant melanoma skin cancer, papillary thyroid / follicular carcinoma, cervical carcinoma in situ, contralateral non-invasive breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2032-07-15 (Estimated); Study Completion 2032-07-15 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  From date of enrollment until to the first recurrence in the ipsilateral breast or chestwall, the regional nodal area, or a distant site or death due to any cause

SECONDARY OUTCOMES:
Overall survival | 5 years
  From date of enrollment until the date of death from any cause.
Distant metastasis-free survival | 5 years
  The time of randomization to the first recurrence in a distant site.
Local-regional recurrence-free survival | 5 years
  The time of randomization to the first recurrence in the ipsilateral breast or chest wall and the regional nodal area.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yang, M.S, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No